CLINICAL TRIAL: NCT03778632
Title: Integration of Individualized Variables of School-age Children Who Stutter Into Intensive Stuttering Group Therapy and the Effect of Emotional Reactivity on Therapy Outcomes
Brief Title: Intensive Stuttering Group Therapy for School-age Children and the Effect of Emotional Reactivity on Therapy Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ilkem Kara, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/621-15
Record Dates: First submitted 2018-12-09; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Stuttering, Childhood; Emotion, Expressed
Keywords: Stuttering; School-age; Emotional reactivity; Wearable technology
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Intensive stuttering group therapy which was included individualized desensitization exercises was applied with the study group. Family training was applied with the parents a month before the therapy. Ten days (4.5 hours a day, a total of 45 hours therapy) of intensive stuttering group therapy was applied.
  Interventions: Behavioral: individualized desensitization exercises
- Control Group (Active Comparator): Standard intensive stuttering group therapy was applied with the control group. Family training was applied with the parents a month before the therapy. Ten days (4.5 hours a day, a total of 45 hours therapy) of intensive stuttering group therapy was applied.
  Interventions: Behavioral: individualized desensitization exercises

INTERVENTIONS:
Behavioral: individualized desensitization exercises — implementing individualized desensitization exercises in standard application of intensive stuttering group therapy for school-age children who stutter

SUMMARY:
The primary objectives of this investigation were two-fold: 1) to investigate whether implementation of individualized desensitization exercises in an intensive stuttering group therapy for school-age children who stutter is superior to the standard application of intensive stuttering group therapy, 2) to examine the relationship between exhibited emotional reactivity (positive and negative affect) and stuttering recovery rates. Secondary objectives included: 1) investigating whether cognitive, affective, linguistic and social scores differ with treatment and, 2) heart rate and skin conductance changes associated with the stuttered utterance during intensive stuttering group therapy activities.

Twelve children (8 to 12 years of age, with equal randomization [1:1]) randomized to two groups; 1) Study group, individualized desensitization exercises implemented in 2 weeks of intensive stuttering group therapy(n=6), 2) Control group, 2 weeks of standard intensive stuttering group therapy(n=6). Children were blinded to treatment arm. The first part of this study was a superiority trial of individualized desensitization exercises in intensive stuttering group therapy. The second part of the study was conducted with the study group during the daily therapy activities of intensive stuttering group therapy to investigate the emotion's effect on therapy outcomes with behavioral and physiological measures.

DETAILED DESCRIPTION:
The investigators hypothesized that (1) implementation of the usage of individualized desensitization exercises in an intensive stuttering group therapy created more effective treatment results than standard implementation of the desensitization exercises in an intensive stuttering group therapy in school-age children who stutter, (2) recovery rates will differ according to exhibited affects before stuttered utterances, (3) heart rate and skin conductivity findings before, during and after the stuttered utterances will differ from the general findings.

Children (n=12) were recruited and randomized in a 1:1 ratio either Control group (n=6) or Study group (n=6) by the study assistant. Randomization was stratified by sex, using a block size of two. For the first part of the study 6 study assessors (speech and language therapy interns who were experienced in the assessment procedure) who were not otherwise involved in the study, were participated in baseline and follow-up assessments. Children were blinded to treatment arm. Video recordings of assessments of the Turkish version of Stuttering Severity Scale-4 were made. Offline assessments of the stuttering severity were done by two research assistants. One of the research assistants was blinded to group assignment and was not otherwise involved in the studies. Video recordings of assessments were labeled by decimal numbers randomly. The masking of the data was done by the study assistant. The second part of the investigation conducted with children in the study group.

For the first part of the study, intervention and family training was applied by a professional therapist who has 7 years of experience in stuttering therapy. When children applied for the baseline assessments, parent training was applied. Training included; (a) general information on stuttering, (b) underlying facts, and (c) how to communicate with their children. At the training session, parents were given an information brochure for teachers of their child. Family training was conducted a month before intensive stuttering group therapy.

The intervention used a hybrid approach which was combined with the evidence-based techniques: speech reconstruction includes fluency shaping and stuttering modification; cognitive restructuring; emotional restructuring; desensitization; video self-modeling.

Standard therapy application included 7 components:

1. Recognition: Speech mechanism, stuttering, fluency or stuttering modification technic, emotions, thoughts, bodily actions, behaviors etc. What is it? Where/When/How to use? Transferring the rationale of the exercise to the participants.
2. Desensitization: It is the process of gradually exposing the participants to the stuttering induced situations (in which there is a negative and very positive mood) by first determining the stuttering induced situations (anxiety ladder exercise used, to begin with). Problem-solving exercises and role-model exercises applied.
3. Technic usage:

   1. Video-model had prepared for fluency shaping which includes easy start, light articulatory contacts, connection, and pausing techniques. At first video model had been watched for once; than clinician asked the children to identify the speech characteristics and they watched the video-model again, chorus readings were done altogether with the clinician and the group, clinician's help retracted gradually and children read the passages alone.
   2. To generalize the fluency technique into speech gradual increase method was used; one-word production games, two-word production games, sentence production games, conversation activities, reading aloud activities, role-model activities were used.
   3. For stuttering modification pull-out technique was introduced during daily activities.
4. Diversified Technic Usage: The skills learned have been used in complex tasks. For example; Making presentations in front of the group and answering questions.
5. Problem-Solving Skills: Identifying problem situations, tagging the emotions, brainstorming, decision making, role-modeling.
6. Generalization: In order to generalize the learned skills to the daily activities, outside of the therapy room, orienteering activity was organized with the adults they hadn't met before. Each child completed a set of tasks outside of the therapy room. Presentation in front of a group of adults (their parents) was organized.
7. Maintenance: In order to maintain the skills gained in therapy after therapy, video self-modeling technique was used. On the last day of therapy, each subject was visually fluent during free speech and reading tasks and was asked to watch these videos every day after therapy.

For both groups of children, desensitization exercises were conducted. Standard intensive stuttering group therapy was applied to the control group while in the study group, clinician's observation was included in the intervention process. Predetermined stuttering inducing situation's table was prepared for each participant. The scenario table was included 5 situations. Clinician observed the children and marked the situations which increased their stuttering. Mostly marked situations were identified for each child. At the end of the first-week children were given instructions for the second week of the therapy. For example; if the child's stuttering severity increased during reading aloud in front of the group, the intensity of the reading-aloud in front of the group exercises was increased for him/her. They were informed that all of them would have special tasks.

Stuttering severity and cognitive, affective, linguistic and social score measures were done 5 times; 1) one month before the therapy, 2) on the first day of the therapy, 3) on the last day of the therapy, 4) one month after the therapy, and 5) three months after the therapy.

For the second part of the study, the images required for the Emotion Facial Action Coding System analysis were recorded during the therapy through CH_TECH SONY CHIPSET 2 MEGAPIXEL IP cameras. A total of six cameras were placed in the therapy room. The analysis of the facial action coding system was carried out by a certified researcher. Increased stuttering moments of subjects in the study group were detected by monitoring and transcription of the camera and microphone recordings at the end of the day. During the time before the fluency technique was thought to the subjects, 10 stuttering moments were identified and the 5-second window before the moment of stuttering was coded.

The evaluations were classified in 2 groups, positive or negative affect. Facial expressions which are expressions specified as non-encoded in Emotion Facial Action Coding System are identified as neutral facial expressions. Positive affect codings were done via observation of facial expressions; AU 12 (extraction of the lip corner) and AU 6 +12 (cheek up with the extraction of the lip corner). Positive affect may be accompanied by AU1 + 2 (eyebrow elevation), AU25 (mouth opening) or AU 26 (loosening of the jaw) (33). If AU12 occurs without AU6, AU12 should occur at least C severity in the intensity classification from 5 to Likert type A to E If AU12 is present with AU6, the intensity of AU12 is B 109, 139. For the coding of negative affects; AU 9 (nose creasing); AU 10 (upper lip elevation); AU 14 (pitting); AU 15 (depression of the lip corner); It is necessary that at least one of the codes AU 20 (lips stretching) and AU 1 + 4 (lifting the eyebrows to the midline and approaching) occur at intensity B.

Skin conductivity and heart rate recordings of participants in the study group were obtained via E4 wristbands. The wristbands were tested on both wrists during the therapy of the control group. As the non-dominant hand wrist's recordings resulted with lower noise levels, the wristbands were worn on the non-dominant side. For the analysis of skin conductivity; 1) online version of EDA-Explorer, 2) Ledalab and 3) Matlab was used. For the heart rate analysis, Matlab was used.

ELIGIBILITY:
Inclusion Criteria:

* very mild to moderate stuttering based on Stuttering Severity Instrument-4-Turkish Version
* no history of intellectual, emotional, academic, hearing, neurological, physiological problems based on parental report
* no history of speech and/or language problems other than stuttering
* not to be received stuttering therapy during the previous six months.

Exclusion Criteria:

-

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
The stuttering severity | One month before therapy to three months after therapy
  Comparison of control group and study group by Turkish version of Stuttering Severity Instrument-4 score change.Stuttering Severity Instrument-4 is an instrument that measures stuttering severity of children in the age range of 6 to16 years. This instrument measures stuttering severity by 3 sub-items; 1)frequency, 2)duration, and 3)physical concominants. evaluates speech naturalness of the children's speech. Lowest available score on this instrument is 6 and is equivalent to very mild stuttering and 36& higher points are equivalent to very severe stuttering.
Emotional reactivity (positive and negative affect) effect on therapy outcome | Collected during first 3 days of the intensive stuttering group therapy to compare the therapy outcomes
  Obtained by means coding behavioral analysis of positive and negative affect. Emotion facial action coding was used to code positive and negative affects. Positive affect coded when the following action units(AU) appeared; AU 12 (extraction of the lip corner) and AU 6 +12 (cheek up with the extraction of the lip corner). Positive affect may be accompanied by AU1 + 2 (eyebrow elevation), AU25 (mouth opening) or AU 26 (loosening of jaw). If AU12 occurs without AU6, AU12 should occur at least C severity in the intensity classification from 5 to likert type A to E If AU12 is present with AU6, the intensity of AU12 is B. For the acceptance of affect as negative; AU 9 (nose creasing); AU 10 (upper lip elevation); AU 14 (pitting); AU 15 (depression of the lip corner); it is necessary that at least one of the codes AU 20 (lips stretching) and AU 1 + 4 (lifting the eyebrows to the midline and approaching) occur at intensity B.

SECONDARY OUTCOMES:
Changes in cognitive, affective, linguistic and social scores | One month before therapy to three months after therapy
  Cognitive, Affective, Linguistic, Motor and Social Rating Scale for School children who stutter is a tool to assess 5 components; 1) cognitive, 2) affective, 3) linguistic, 4) motor, and 5) social. Cognitive component assess the child's awareness, knowledge understanding of stuttering. The affective component gives information on the child's feelings/attitudes related to stuttering & positive/negative attributes of him/her self. The linguistic component assess: overall language, speech sound & vocabulary abilities and, stuttering with regards to the length and complexity of utterances. The social component assess the child's approach to the social situations. At the end every component was rated on a scale of 1-5 (1= low concern, 5= high concern).
Heart rate changes | Collected during first 3 days of the intensive stuttering group therapy
  Obtained via wearable technology. The average of general heart rate values which were expressed in beat per minute was compared with the average heart rate values occurred in one-minute window before and after the stuttered utterances.
Skin conductance changes | Collected during first 3 days of the intensive stuttering group therapy
  Obtained via wearable technology. The average general of skin conductivity values which were expressed in microsiemens was compared with the average skin conductivity values occurred in one-minute window before and after the stuttered utterances.

CONTACTS AND LOCATIONS:
Overall Officials: Mavis Emel Kulak Kayikci, Assoc. Prof., Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF